CLINICAL TRIAL: NCT01178489
Title: Recovery at the Post Anaesthetic Care Unit After Fast-track Hip and Knee Arthroplasty
Brief Title: Recovery at the Post Anaesthetic Care Unit After Hip and Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Other Study IDs: H-1-2010-FSP
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: PACU Stay After THA Under Spinal Anaesthesia; PACU Stay After TKA Under Spinal Anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing arthroplasty: Patients undergoing primary, unilateral, total hip or knee arthroplasty under spinal anaesthesia

SUMMARY:
To clarify patient related problems in the Post Anaesthetic Care Unit (PACU) immediately after fast-track hip and knee arthroplasty.

DETAILED DESCRIPTION:
In this prospective, consecutive, observational cohort study we examine:

1. Patient related problems in the PACU after hip and knee arthroplasty simply to answer the question "Why in PACU?", using a modified version of the national guidelines for patient observation in PACU.
2. The time spent in PACU with the modified version of the national guidelines for patient observation in PACU.
3. If the modified version of the national guidelines for patient observation in PACU results in patient related problems in the ward afterwards.

ELIGIBILITY:
Inclusion Criteria:

* primary, unilateral, total hip or knee arthroplasty by one of three surgeons using the same technique, and under spinal anaesthesia

Exclusion Criteria:

* Bilateral arthroplasty
* Revision arthroplasty
* General anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary, unilateral, total hip or knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time to meet PACU discharge criteria | 3 hours

SECONDARY OUTCOMES:
Actual discharge time from PACU | 3 hours
Clinical and logistic factors detaining patients in PACU | 3 hours
Potential complications at the surgical ward | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Troels H Lunn, M.D., Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark